CLINICAL TRIAL: NCT02845336
Title: An Open Label Trial of Celecoxib in the Treatment of Mild Thyroid Eye Disease
Brief Title: Celecoxib for Thyroid Eye Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00094787
Record Dates: First submitted 2016-07-20; First posted 2016-07-27 (Estimated); Results first posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Celecoxib; Lubricant Eye Drops

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Celecoxib (Experimental): Patients who are randomized to treatment with celecoxib 100mg pills by mouth twice a day for 3 months, in addition to standard of care treatment as described under the Control arm
  Interventions: Drug: Celecoxib; Drug: artificial tears
- Control (Active Comparator): Patients who are randomized to standard treatment (requiring no prescription medication, but standard recommendations such as artificial tears, avoiding cigarette smoke)
  Interventions: Drug: artificial tears

INTERVENTIONS:
Drug: Celecoxib — celecoxib 100mg PO twice per day for 3 months
  Other Names: Celebrex
  Arms: Celecoxib
Drug: artificial tears — Standard care for mild thyroid eye disease is lubrication with artificial tears (over the counter), avoidance of cigarette smoke.

SUMMARY:
Thyroid eye disease (TED) is an autoimmune disorder in which the immune system attacks orbital tissues, resulting in characteristic changes in eyelid position, globe position in the orbit, extraocular muscle balance, and optic nerve function. TED is a potentially blinding disease, and current treatments largely consist of nonspecific reduction of inflammation using corticosteroids or radiation therapy. Regardless of treatment, once TED progresses from its inflammatory phase to a more fibrotic, resolution phase, the orbital changes become fixed and can be modified only by surgery.

The investigators propose to treat a cohort of patients with active TED using a selective COX-2 inhibitor, celecoxib, and to compare these patients to an observational control group. The investigators hypothesize that celecoxib will reduce the severity of disease and/or prevent progression to proptosis, diplopia, and corneal exposure or compressive optic neuropathy.

DETAILED DESCRIPTION:
The investigators intend to use celecoxib, a non-steroidal anti-inflammatory drug approved by the Food and Drug Administration (FDA) for the treatment of pain, osteoarthritis, rheumatoid arthritis, and ankylosing spondylitis, as a treatment for active TED. In vitro data have shown that transformation of orbital fibroblasts into adipocytes is mediated by cyclooxygenase-2 (COX-2), and a case report suggests that COX-2 inhibition can improve TED in the acute phase. Thus, the investigators intend to evaluate the efficacy of COX-2 inhibition in the treatment of active TED and its ability to improve both the acute inflammatory signs and more permanent fibrotic changes of quiescent disease. The investigators will enroll patients with active TED and treat them for 3 months (a characteristic period of disease activity) and compare this to standard treatments for mild active TED (observation, with over the counter interventions such as lubrication with artificial tears) to assess efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Recent diagnosis of thyroid eye disease (within the past 3 months)
* Have ocular symptoms or signs of TED with a clinical activity score (CAS) of at least 3

Exclusion Criteria:

* Pregnancy
* Previous treatment with corticosteroid for TED for >2wks
* Previous treatment with orbital radiation for TED
* Impaired renal function
* Impaired hepatic function
* Treatment with antihypertensive medications except beta-blockers
* History of congestive heart failure, cardiac valvular disease, or coronary artery disease
* Allergy to NSAID or previous adverse reaction (ie. GI bleeding)
* Vision loss due to compressive optic neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-03-05 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J McCulley, MD, Principal Investigator — Wilmer Eye Institute, Johns Hopkins School of Medicine
Locations (1):
- Wilmer Eye Institute, Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Celecoxib | Control
Started | 6 | 1
Completed | 1 | 0
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Inability to get medication | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib | Control | Total
Number analyzed (Participants) | 6 | 1 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 1 | 6
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 2 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Thyroid Eye Disease Clinical Activity Score
Description: A clinical score based on examination findings at each clinic visit. Clinical Activity Scores ranged from 0 to 10; 0 = Normal 1-3 = Mild 4-6 = Moderate 7-10 = Severe
Time Frame: At baseline, 1, 3 and 6 months
Population: No participant in control arm was assessed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib | Control
Number analyzed (Participants) | 1 | 0
Participants
  Baseline: Normal | 0 |
  Baseline: Mild | 0 |
  Baseline: Moderate | 1 |
  Baseline: Severe | 0 |
  1 month: Normal | 0 |
  1 month: Mild | 0 |
  1 month: Moderate | 1 |
  1 month: Severe | 0 |
  3 months: Normal | 0 |
  3 months: Mild | 0 |
  3 months: Moderate | 1 |
  3 months: Severe | 0 |
  6 months: Normal | 0 |
  6 months: Mild | 0 |
  6 months: Moderate | 1 |
  6 months: Severe | 0 |

2. Secondary Outcome: Proptosis as Measured in Millimeters With an Exophthalmometer (Right Eye)
Description: A clinical measure of how prominent the eyes are and any change in this measure over the duration of the study, as measured in millimeters with an exophthalmometer.
Time Frame: At baseline, 1, 3 and 6 months
Population: No participant in control arm was assessed for this outcome measure.
Measure: Number; unit: millimeters
Arm/Group | Celecoxib | Control
Number analyzed (Participants) | 1 | 0
millimeters
  Baseline | 20.5 |
  1 month | 20.5 |
  3 months | 20.5 |
  6 months | 20.5 |

3. Secondary Outcome: Proptosis as Measured in Millimeters With an Exophthalmometer (Left Eye)
Description: as for outcome 2
Time Frame: At baseline, 1, 3 and 6 months
Population: No participant in control arm was assessed for this outcome measure.
Measure: Number; unit: millimeters
Arm/Group | Celecoxib | Control
Number analyzed (Participants) | 1 | 0
millimeters
  Baseline | 21.5 |
  1 month | 21.5 |
  3 months | 21.5 |
  6 months | 21.5 |

4. Secondary Outcome: Number of Participants With Ocular Misalignment
Description: Presence or absence of ocular misalignment measured in prism diopters.
Time Frame: At baseline
Population: No participant in control arm was assessed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib | Control
Number analyzed (Participants) | 1 | 0
Participants
  Present | 0 |
  Absent | 1 |

5. Secondary Outcome: Number of Participants With Ocular Misalignment
Description: Presence or absence of ocular misalignment measured in prism diopters.
Time Frame: At 1 month
Population: No participant in control arm was assessed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib | Control
Number analyzed (Participants) | 1 | 0
Participants
  Present | 0 |
  Absent | 1 |

6. Secondary Outcome: Number of Participants With Ocular Misalignment
Description: Presence or absence of ocular misalignment measured in prism diopters.
Time Frame: At 3 months
Population: No participant in control arm was assessed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib | Control
Number analyzed (Participants) | 1 | 0
Participants
  Present | 0 |
  Absent | 1 |

7. Secondary Outcome: Number of Participants With Ocular Misalignment
Description: Presence or absence of ocular misalignment measured in prism diopters.
Time Frame: At 6 months
Population: No participant in control arm was assessed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib | Control
Number analyzed (Participants) | 1 | 0
Participants
  Present | 0 |
  Absent | 1 |

8. Secondary Outcome: Eyelid Retraction as Measured in Millimeters (Right Eye)
Description: A clinical measure of the most common manifestation of thyroid eye disease--change in eyelid retraction as measured in millimeters at each visit over the duration of the study.
Time Frame: At baseline, 1, 3 and 6 months
Population: No participant in control arm was assessed for this outcome measure.
Measure: Number; unit: millimeters
Arm/Group | Celecoxib | Control
Number analyzed (Participants) | 1 | 0
millimeters
  Baseline | 0.5 |
  1 month | 0.5 |
  3 months | 0.5 |
  6 months | 0.5 |

9. Secondary Outcome: Eyelid Retraction as Measured in Millimeters (Left Eye)
Description: as for outcome 8
Time Frame: At baseline, 1, 3 and 6 months
Population: No participant in control arm was assessed for this outcome measure.
Measure: Number; unit: millimeters
Arm/Group | Celecoxib | Control
Number analyzed (Participants) | 1 | 0
millimeters
  Baseline | 2 |
  1 month | 2 |
  3 months | 2 |
  6 months | 2 |

10. Secondary Outcome: Quality of Life as Assessed by a Thyroid Eye Disease Specific Survey of Quality of Life
Description: Thyroid eye disease specific survey of quality of life will be administered, and change in quality of life score over the duration of the study will be measured.
Time Frame: 6 months
Population: This measure was not assessed. No data was collected.
Arm/Group | Celecoxib | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: No participant enrolled in the control arm was followed for adverse events. Only 1 participant in the treatment arm was followed for adverse events. The rest were either lost to follow up or didn't get medication.
Arm/Group | Celecoxib | Control
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT02845336/Prot_SAP_000.pdf